CLINICAL TRIAL: NCT01169506
Title: A New Method of Sublingual Tonometry to Assess Tissue Perfusion in Patients With COPD and Healthy Individuals
Brief Title: Sublingual Tonometry to Assess Tissue Perfusion in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Acronym: subton
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Attila Somfay, MD, PhD, Department of Pulmonology, University of Szeged, Hngary
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: nagymaci54
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2009-03

CONDITIONS: COPD; Healthy Subjects
Keywords: blood gas analysis; ventilatory insufficiency
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD patients and healthy individuals (Experimental)
  Interventions: Device: sublingual silicon capillary

INTERVENTIONS:
Device: sublingual silicon capillary — Stable patients with COPD and healthy individuals were asked to open their mouth and a small butterfly silicon capillary was placed sublingually. After 15 minutes, while the mouth was closed completely and nose breathing was performed, the capillary system was connected to a capnometer and sublingual tonometric PCO2 was measured. At the same time, PETCO2 was also measured and arterial blood was drawn for pH, PO2 and PCO2 analysis
  Other Names: sublingual tonometry, tissue perfusion, ventilation

SUMMARY:
Sublingual positioning of a silicon capillary system is applied. After 15 min, while the individual is in resting position with closed mouth and normal tidal breathing through the nose is performed, the silicon capillary system is connected to a capnometer and CO2 tension is measured.

The investigators hypothesis is that this setup offers a non-invasive assessment of ventilatory efficiency with similar accuracy as arterial PCO2.

DETAILED DESCRIPTION:
We have developed a new silicon capillary system for sublingual monitoring of CO2 tension in order to assess tissue perfusion. This set up is non-invasive, cheaper than previous tonometry devices and easier to apply in clinical routine. We have recruited patients with stable COPD and healthy individuals.

Sublingual tonometry results were evaluated after 15 min of tidal breathing with a capnometer for CO2 tension. Corresponding end tidal CO2 (PETCO2)and arterial blood gas values (pH, PaCO2, PaCO2) were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with stable disease

Exclusion Criteria:

* acute exacerbation of COPD

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
sublingual tonometric PCO2 - arterial PCO2 | one year

SECONDARY OUTCOMES:
sublingual tonometric PCO2 - PETCO2 | one year

CONTACTS AND LOCATIONS:
Overall Officials: Attila Somfay, MD,PhD, Principal Investigator — Department of Pulmonology, University of Szeged, Hungary
Locations (1):
- Department of Pulmonology, Albert Szent-Györgyi Clinical Center, University of Szeged, Deszk, Hungary

REFERENCES:
- [Background] Boda D, Kaszaki J, Talosi G. A new simple tool for tonometric determination of the PCO2 in the gastrointestinal tract: in vitro and in vivo validation studies. Eur J Anaesthesiol. 2006 Aug;23(8):680-5. doi: 10.1017/S026502150600055X. PMID 16805933